CLINICAL TRIAL: NCT04364919
Title: Effects of Aerobic Exercise on Sleep Quality and Maternal-fetal Attachment in Pregnant Women: A Randomized Controlled Pilot Study
Brief Title: Aerobic Exercise on Prenatal Sleep Quality and Maternal-fetal Attachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chung-Hey Chen, Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSC102-2314-B006-063-MY2
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Effects of Aerobic Exercise in Pregnant Women
Keywords: aerobic exercise; prenatal care; sleep quality; maternal-fetal attachment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: In addition to routine care, the experimental group was given a DVD and instructed to engage in the aerobic exercise program shown on the DVD. The DVD with low-impact aerobic exercises developed by the researchers in collaboration with a qualified prenatal yoga teacher. The program incorporated modified yoga movements suitable for pregnant women. Women in experimental group were instructed to use the DVD 3 times a week for 3 months. The control group received routine prenatal care only.
Who Masked: Participant
Masking Description: One hundred and forty women who met the inclusion criteria and returned their consent documents were systematically assigned, from a random starting point to experimental (n = 70) or a control (n = 70) group. Women usually talk to each other during the prenatal check and this could cause study data contamination, so we used a month as the unit of allocation to avoid between-group data contamination. The first month collecting data was control group decided by drawing lots (two lots which were marked "E" for experimental group and marked "C" for control group in a sack). Research assistant drew the lot from the sack. Then, the following month, group allotment was systematically assigned in sequence to either the experimental group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercise intervention (Experimental): The intervention group received a DVD with low-impact aerobic exercises developed by the researchers in collaboration with a qualified prenatal yoga teacher. With a soft musical background, the exercise actions were arranged in following order: warm-up → neck → shoulder → arm → chest → waist →leg → regulating the breathing. The first 14.5 minutes of the yoga exercises were performed in a sitting position, followed by 3.5 minutes in standing position, and then returning to 2 minutes in sitting position. The exercise program requires twenty minutes to complete. Women were instructed to use the DVD 3 times a week for 3 months.
  Interventions: Behavioral: aerobic exercise program
- control group (No Intervention): The control group received routine prenatal care only.

INTERVENTIONS:
Behavioral: aerobic exercise program — The program incorporated modified yoga movements suitable for pregnant women. The DVD provides an illustration with the written caption, "Please take enough water before exercise, and wear loose and comfortable clothes in a suitable environment. If you feel tired, stop exercising immediately." The DVD's narrator then says, "Now you are ready to prepare a comfortable, solid chair with a chair back." With a soft musical background, the exercise actions were arranged in following order: warm-up → neck → shoulder → arm → chest → waist →leg → regulating the breathing. The first 14.5 minutes of the yoga exercises were performed in a sitting position, followed by 3.5 minutes in standing position, and then returning to 2 minutes in sitting position. The exercises were developed as a progressive program in order to achieve the goals of strength-conditioning, moderate-intensity exercise (ACOG, 2015).
  Arms: aerobic exercise intervention

SUMMARY:
A growing body of evidence suggests that exercise is an important contributor to maternal health and is beneficial to infants. A single-blinded randomised experimental study was used to evaluate the effect of aerobic exercise on sleep quality and maternal-fetal attachment in pregnancy women. 140 eligible pregnant women were systematically assigned, with a random start to experimental group (n = 70) received a 20 minutes aerobic exercise video and was instructed to exercise at least three times a week for 3 months at home, while the control group (n = 70) received the usual care only. The Pittsburgh Sleep Quality Index and Modified Maternal-Fetal Attachment Scale were used to assess outcomes measured before the intervention and at 4 and 12 weeks postintervention. Paired sample t-tests were conducted before and after aerobic exercise to measure whether there were any statistically significant changes in outcome variables.

DETAILED DESCRIPTION:
3.1 | Study design In this study, a single-blinded, randomized, controlled trial with a prospective pretest-posttest experimental design was implemented to examine the effects of low-impact aerobic exercise with modified yoga movements on sleep quality and maternal-fetal attachment in pregnant women.

3.2 | Participants Participants for this study were recruited from the prenatal clinic of a medical center in southern Taiwan. A sample size of 63 per group was considered sufficient to estimate a medium effect of .50 with α-value of 0.05 and a power of 0.08 (Polit & Beck, 2011). Considering a 20% attrition rate over 3 months, 140 pregnant women were enrolled.

3.3 | Intervention The intervention group received a DVD with low-impact aerobic exercises developed by the researchers in collaboration with a qualified prenatal yoga teacher. The program incorporated modified yoga movements suitable for pregnant women. The DVD provides an illustration with the written caption, "Please take enough water before exercise, and wear loose and comfortable clothes in a suitable environment. If you feel tired, stop exercising immediately." The DVD's narrator then says, "Now you are ready to prepare a comfortable, solid chair with a chair back." With a soft musical background, the exercise actions were arranged in following order: warm-up → neck → shoulder → arm → chest → waist →leg → regulating the breathing. The first 14.5 minutes of the yoga exercises were performed in a sitting position, followed by 3.5 minutes in standing position, and then returning to 2 minutes in sitting position. The exercises were developed as a progressive program in order to achieve the goals of strength-conditioning, moderate-intensity exercise (ACOG, 2015). The yoga teacher instructed the participants to touch their heart with their right hand and their abdomen with their left hand, feeling a connection with the fetus in the warm-up and in the final breath-regulating stage of exercise (2 minutes). An expert video producer edited the DVD for sound, animation, and subtitles. The exercise program requires twenty minutes to complete. Women were instructed to use the DVD 3 times a week for 3 months. The DVD was reviewed for content validity by two clinical obstetric nursing experts, and in addition, two pregnant women in their second trimester reviewed the DVD for face validity.

3.5 | Procedure and ethical considerations The present study was carried out from January to October 2014 after approval was obtained from the institutional review board of the participating institution. One hundred and forty women who met the inclusion criteria and returned their consent documents were systematically assigned, from a random starting point to experimental (n = 70) or a control (n = 70) group. Women usually talk to each other during the prenatal check and this could cause study data contamination, so we used a month as the unit of allocation to avoid between-group data contamination. The first month collecting data was control group decided by drawing lots (two lots which were marked "E" for experimental group and marked "C" for control group in a sack). Research assistant drew the lot from the sack. Then, the following month, group allotment was systematically assigned in sequence to either the experimental group or the control group.

In addition to routine care, the experimental group was given the DVD and instructed to engage in the aerobic exercise program shown on the DVD. The control group received routine prenatal care only. The two groups were asked to complete the demographic data form, the MMFAS, and the PSQI at 3 time periods: before the intervention, at 4 weeks, and 12 weeks post-intervention. All participants in both groups received a small gift after completing the pretests. The latter two sets of questionnaires were mailed with postage-paid, pre-addressed envelopes to all of the participants for them to complete and return. Sixty-one participants in the experimental group and 62 participants in the control group completed the 1-month posttests; 51 participants in the experimental group and 47 participants in control group completed the 3-month posttests. The CONSORT diagram of this study is shown in Figure 1. The experimental group participants were asked to complete an open-ended question on the subjective benefits of practicing aerobic exercise.

3.6 | Data analysis Tests for differences in baseline characteristics between the two groups included the χ2 test for categorical variables and the t-test for continuous variables. The effectiveness of yoga-based low-impact aerobic exercise on maternal-infant attachment and sleep quality was determined by a paired t-test. All results with p < .05 were considered statistically significant. The SPSS (version 17.0 for Windows, SPSS Inc., Chicago, IL, USA) statistical software package was used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were (a) uncomplicated pregnancy, (b) between 16 and 30 weeks gestation, and (c) informed consent to participate.

Exclusion Criteria:

* Women were excluded if they reported any contraindications to aerobic exercise during pregnancy according to the 2015 ACOG guidelines.

Ages: 23 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) was used to measure subjective sleep quality during pregnancy. The PSQI, developed by Buysse et al. (1989), contains 19 items and measures 7 components of sleep quality, including habitual sleep efficiency, sleep latency, sleep duration, sleep disturbances, use of sleep medication, daytime dysfunction, and subjective sleep quality. Each component is evaluated on a 4-point Likert scale, with 0 representing better sleep and 3 representing worse sleep. The summed scores range from 0 to 21, with scores over 5 indicating poor sleep quality and scores less than or equal to 5 indicating good sleep quality.
Modified Maternal-Fetal Attachment Scale | 12 weeks
  The Modified Maternal-Fetal Attachment Scale (MMFAS) was used to measure maternal attachment to the fetus. The MMFAS was developed by merging the Muller's (1993) Prenatal Attachment Inventory with the Cranley's (1981) Maternal-Fetal Attachment Scale. The MMFAS Mandarin language version comprises 39 items addressing four factors: interacting with the fetus, giving of self, identifying the fetus, and fantasizing (Hsu & Chen, 2001). Each item is ranked on a 5-point Likert scale, with 0 = never and 4 = always. Scores range from 0 to 156, with higher scores indicating greater maternal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hey Chen, PhD, Principal Investigator — College of Medicine, National Cheng-Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No